CLINICAL TRIAL: NCT03918811
Title: Comparison of Two Extubation Techniques in Critically Ill Adult Patients (ExtubAR Trial): Randomized Clinical Trial
Brief Title: Comparison of Two Extubation Techniques in Critically Ill Adult Patients
Acronym: ExtubAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the outbreak of the SARS-CoV-2 pandemic in Argentina and the lack of information about the potential risks of contamination from extubation and aerosolization, we stopped recruiting patients before achieving the predefined sample size.
Sponsor: Hospital Donación Francisco Santojanni (Other)
Collaborators: Matías Bertozzi (Unknown); Marco Bezzi (Unknown); Borello, Silvina, M.D. (Individual); Daniela Castro (Unknown); Victoria Di Giorgio (Unknown); Mariana Aguirre (Unknown); Karina Miralles (Unknown); Diego Noval (Unknown); Sebastián Fredes (Unknown); Eliana Wilhelm (Ambiguous); Mauricio Zakimchuk (Unknown); Julián Buffarini Cignoli (Unknown); Mariana Bernardini (Unknown); Leticia Rey (Unknown); Valeria Pieroni (Unknown); Pablo D´Annunzio (Unknown); Gustavo Plotnikow (Unknown); Romina Prato (Unknown); Matías Lompizano (Unknown); María Guaymas (Unknown); Matías Accoce (Unknown); Javier Dorado (Unknown); Gimena Cardoso (Unknown); Patricia Torres (Unknown); Vanesa Pavlotsky (Unknown); Emiliano Navarro (Ambiguous); Eliana Markman (Ambiguous); Paula Di Nardo (Unknown); Ivonne Kunzi Steyer (Unknown); Thomsen, Carolina, M.D. (Individual); Cecilia Palacios (Unknown); Mariela Davies (Unknown); Mercedes Ruffo (Unknown); Victoria Leon (Unknown); Fernando Tapia (Unknown)
Responsible Party: Principal Investigator, Mauro Andreu, Physical Therapist, Hospital Donación Francisco Santojanni
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-2018-05
Record Dates: First submitted 2019-04-14; First posted 2019-04-18 (Actual); Results first posted 2021-02-09 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-01

CONDITIONS: Weaning Failure; Mechanical Ventilation Complication
Keywords: airway extubation; extubation methods; positive pressure; positive-pressure extubation; tracheal extubation; positive-pressure ventilation; extubation complications

STUDY DESIGN:
Intervention Model Description: superiority
Who Masked: Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, blinding of the subject and the operators responsible for extubation is not possible. The person in charge of data statistical analysis and the evaluator who assess and record outcome measures will be blinded to the allocated intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Pressure Extubation Technique (Experimental): ETT is removed in PSV 15/10 mode and without endotracheal suction.
  Interventions: Procedure: Positive Pressure Extubation Technique
- Traditional Extubation Technique (Active Comparator): ETT is removed with continuous endotracheal suction
  Interventions: Procedure: Traditional Extubation Technique

INTERVENTIONS:
Procedure: Positive Pressure Extubation Technique — Positive-pressure extubation is performed by only one operator. Ventilator parameters are set to pressure support ventilation mode, with an inspiratory pressure of 15 cm H2O and PEEP of 10 cm H2O. Then, the cuff is deflated, and the ETT is removed without endotracheal suction. Once the ETT is removed, a suction catheter is introduced through the mouth to suction secretions drawn to the oropharynx by the air flow from the ventilator passing between the ETT and the larynx.
  Arms: Positive Pressure Extubation Technique
Procedure: Traditional Extubation Technique — Traditional extubation is performed by 2 operators. Without reconnection to the ventilator, the closed suction system catheter is introduced by one of the operators into the ETT and suctioning is initiated. The cuff is immediately deflated by the other operator, and the ETT is removed with continuous endotracheal suction during the whole procedure by the first operator.
  Arms: Traditional Extubation Technique

SUMMARY:
Orotracheal extubation consists in the removal of the endotracheal tube (ETT) when it is no longer required. This procedure may carry a considerable risk of complications and extubation failure. The literature points out two methods of extubation: the traditional method and the positive pressure method.

In a noninferiority clinical trial it was demonstrated that EOT with positive pressure and without endotracheal suction was a safe technique and could be better than traditional extubation. Although prior studies reported better clinical outcomes with the positive pressure extubation technique, its superiority has not been deeply studied yet. Therefore, the objective of our study is to determine whether the positive pressure OTE technique, compared with the traditional OTE technique, reduces the incidence of major postextubation complications (up to 60 minutes) in critically ill adult patients.

DETAILED DESCRIPTION:
Design: Multicenter randomized controlled clinical trial Methods: Critically ill adult subjects on invasive mechanical ventilation who met extubation criteria will be included. Will be randomly assigned to positive-pressure extubation (n=389) or to traditional extubation (n=389).

The main variable will be incidence of major complications.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Invasive mechanical ventilation through an endotracheal tube,
* Successfully complete a spontaneous breathing trial
* Adequate level of consciousness (Glasgow Coma Score >8)
* Effective cough.
* Written informed consent from a relative or legal representative.

Exclusion Criteria:

* History of upper airway injury or surgery
* Previously extubated or tracheostomized
* Noninvasive ventilation (NIV) as a weaning method
* Decision to not reanimate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03-26 (Actual); Study Completion 2020-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro F Andreu, Prof, Principal Investigator — Hospital Santojanni
Locations (1):
- Hospital Santojanni, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andreu MF, Salvati IG, Donnianni MC, Ibanez B, Cotignola M, Bezzi M. Effect of applying positive pressure with or without endotracheal suctioning during extubation: a laboratory study. Respir Care. 2014 Dec;59(12):1905-11. doi: 10.4187/respcare.03121. Epub 2014 Nov 25. PMID 25425709
- [Background] Andreu MF, Dotta ME, Bezzi MG, Borello S, Cardoso GP, Dib PC, Garcia Schustereder SL, Galloli AM, Castro DR, Di Giorgio VL, Villalba FJ, Bertozzi MN, Carballo JM, Martin MC, Brovia CC, Pita MC, Pedace MP, De Benedetto MF, Delli Carpini J, Aguirre P, Montero G. Safety of Positive Pressure Extubation Technique. Respir Care. 2019 Aug;64(8):899-907. doi: 10.4187/respcare.06541. Epub 2019 Mar 26. PMID 30914493

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to the ICU, Emergency Unit or Coronary Unit between April 1, 2019, and March 26, 2020, were included in the analysis. We included patients aged > 18 years, requiring invasive mechanical ventilation through an ETT, who had successfully completed a spontaneous breathing trial and met the following OTE criteria: an adequate level of consciousness and effective cough (cough at order and/or at endotracheal suctioning). Informed consent was also required.
Pre-assignment Details: Patients with a history of upper airway (UA) injury or surgery, with a limited therapeutic effort, who had previously been extubated or tracheostomized, or who had required noninvasive mechanical ventilation (NIMV) as a weaning method were excluded from our study. A total of 2567 patients met the eligibility criteria, 1842 were excluded from the study, and 725 were randomly assigned to the traditional extubation group (n=358) and positive pressure extubation group (n=367).
Period: Overall Study
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
Started | 367 | 358
Completed | 363 | 345
Not Completed | 4 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique | Total
Number analyzed (Participants) | 367 | 358 | 725
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 203 | 203 | 406
  >=65 years | 164 | 155 | 319
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 64 [52 to 74] | 63 [51 to 73] | 63 [51 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 134 | 280
  Male | 221 | 224 | 445
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 367 | 358 | 725
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Argentina | 367 | 358 | 725
High Risk of Extubation Failure [Count of Participants; unit: Participants] — High risk of extubation failure was defined as the presence of at least one of the following criteria: age ≥66 years, moderate or severe COPD, >1 comorbidities, body mass index >30, congestive heart failure as main reason from IMV, difficult intubation, IMV >7 days, a requirement of suctioning respiratory secretions (>2 suctions within 4 h before the orotracheal extubation (OTE)), difficult or prolonged weaning and/or APACHE II (Acute Physiology and Chronic Health disease Classification System II) a day before the OTE >12.
  Participants | 302 | 295 | 597

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Major Post Extubation Complications
Description: Clinical evidence of at least one of the following:
  * Upper airway obstruction
  * Desaturation
  * Vomiting
Time Frame: Within15 minutes after extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
Number analyzed (Participants) | 363 | 345
Participants | 89 | 96

2. Secondary Outcome: Number of Participants With Minor Post Extubation Complications
Description: Clinical evidence of at least one of the following:
  * Hypertension
  * Tachycardia
  * Tachypnea
  * Poor respiratory mechanics
  * Bronchospasm
  * Severe cough
  * Post obstructive pulmonary edema
Time Frame: Hypertension, Tachycardia, Tachypnea or Poor Respiratory Mechanics, within 15 minutes after extubation. Bronchospasm, Severe cough or Post Obstructive Pulmonary Edema, within 60 minutes after extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
Number analyzed (Participants) | 363 | 345
Participants | 144 | 156

3. Secondary Outcome: Number of Participants With Overall Post Extubation Complications
Description: Clinical evidence of at least one of the following:
  * Upper airway obstruction
  * Desaturation
  * Vomiting
  * Hypertension
  * Tachycardia
  * Tachypnea
  * Poor respiratory mechanics
  * Bronchospasm
  * Severe cough
  * Post obstructive pulmonary edema
Time Frame: Upper airway obstruction, Desaturation, Vomiting, Hypertension, Tachycardia, Tachypnea, Poor Respiratory Mechanics, within 15 minutes after extubation. Bronchospasm, Severe cough or Post Obstructive Pulmonary Edema, within 60 minutes after extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
Number analyzed (Participants) | 363 | 345
Participants | 190 | 197

4. Secondary Outcome: Number of Participants With Post Extubation Pneumonia
Description: Presence of a new radiographic infiltrate or progression of infiltrates prior to extubation and any of the following: fever, leukocytosis (greater than 10,000 / mm3) or leukopenia (less than 4,000 / mm3) compared to the value prior to extubation and increase in the amount or change in the quality of tracheobronchial secretions.
Time Frame: Within 72 hours after extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
Number analyzed (Participants) | 363 | 345
Participants | 18 | 24

5. Secondary Outcome: Number of Participants With Extubation Failure
Description: Use of Non Invasive Ventilation to treat the failure or need of reintubation.
Time Frame: Within 72 hours after extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
Number analyzed (Participants) | 363 | 345
Participants | 48 | 61

6. Secondary Outcome: Number of Participants That Required Reintubation
Description: Need of reintubation.
Time Frame: Within 72 hours after extubation.
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
Number analyzed (Participants) | 363 | 345
Participants | 44 | 51

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Positive Pressure Extubation Technique | Traditional Extubation Technique
All-Cause Mortality (participants affected / at risk) | 41/363 | 45/345
Serious Adverse Events (participants affected / at risk) | 0/363 | 0/345
Other Adverse Events (participants affected / at risk) | 0/363 | 0/345

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/11/NCT03918811/Prot_SAP_000.pdf